CLINICAL TRIAL: NCT04638413
Title: Cognitive Training Through Gaming and Walking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Sarah Salvy, Professor, Department of Medicine, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00001030
Record Dates: First submitted 2020-10-29; First posted 2020-11-20 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Healthy Lifestyle
MeSH Terms: interventions — Walking

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walking regimen (W) (Experimental)
  Interventions: Behavioral: Walking (W)
- Walking regimen + gamified inhibitory control training (W+PolyRules!) (Experimental)
  Interventions: Behavioral: Walking + PolyRules! (W+PolyRules!)

INTERVENTIONS:
Behavioral: Walking (W) — Participants engage in 30 min of walking daily, for three weeks.
  Arms: Walking regimen (W)
Behavioral: Walking + PolyRules! (W+PolyRules!) — Participants alternate between 30 min of walking on half of the days and 30 min of gamified inhibitory control on the other days.
  Arms: Walking regimen + gamified inhibitory control training (W+PolyRules!)

SUMMARY:
This pilot study evaluated the feasibility of combining daily walking and gamified inhibitory control training. Feasibility was defined by recruitment, retention, and adherence to arm requirements, with secondary, exploratory analyses examining cognitive function outcomes

DETAILED DESCRIPTION:
This pilot study evaluated the feasibility of combining a walking regimen with gamified inhibitory control training (PolyRules!), compared to walking alone, on cognitive outcomes among healthy adults (ages 18 and over). Participants (n=30) will first be asked to wear a Fitbit for one week to capture baseline activity. Participants will then be randomized to (1) walking alone regimen or (2) walking + gamified inhibitory control training for three weeks. Cognitive assessments will be conducted at enrollment and at the end of the 4-week study protocol. The primary outcome of the pilot trial is feasibility as defined by recruitment, retention, and adherence to arm requirements. Engagement and adherence will be operationalized as the frequency and duration of cognitive training passively recorded on the PolyRules! app and frequency and duration of walking as monitored by Fitbit data. Secondary outcomes examined cognitive function outcomes performance: changes in attention and inhibitory control [Cancellation task, Flanker task, and Rule Set task]; And working memory capacity [N-Back task, Letter-Numbers task, and Corsi task]. Qualitative indicators will also be collected via semi-structured interviews to capture participants' satisfaction, perceived benefits of- and/or barriers to engaging with the cognitive training and/or walking regimens.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, write, and speak English with acceptable visual and auditory acuity, as the app is only available in English
* Able and willing to walk independently with or without walking aids
* Able and willing to engage in 30 minutes of walking daily
* Able and willing to wear a fitness tracking device (e.g. Fitbit)
* Not currently engaging in a daily walking regimen of 30 minutes or more a day

Exclusion Criteria:

* Visual impairments that would preclude participants from using the app
* Undergoing active cancer treatment
* Diagnosis of peripheral neuropathy, severe musculoskeletal or neurodegenerative disease (e.g. dementia, multiple sclerosis, Parkinson's disease, Huntington's disease, etc.)
* Taking medications that may affect cognitive function
* Pacemaker, implantable cardiac defibrillator, neuro-stimulation devices, cochlear implants, implantable hearing aids, or other electronic medical equipment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
Recruitment and Retention | Immediately after the 4 week study
  Percentage of randomized participants who complete the final study visit/assessment at the end of the intervention period. Completion is defined as providing primary outcome data (objective adherence logs), calculated as (number completing final assessment / number randomized) × 100.
Rate of walking regimen completion | Daily starting at baseline and for 4 continuous weeks
  Activity will be continuously recorded by the Fitbit to monitor whether participants engage in daily physical activity. There are a total of 9 and 18 walking sessions that may be completed for participants assigned to the control group and intervention group, respectively. Competing one of the sessions entails completing 30 minutes of walking with a wearable. A ratio of completion will be calculated using the number of walking sessions completed over the total amount of sessions possible.
Rate of gamified cognitive training completion | Daily starting at baseline and for 4 continuous weeks
  Participants' interactions with the app (PolyRules!) will be passively recorded by the software to monitor training session completion. There are a total of 8 or more sessions that may be completed for participants assigned to the condition. Competing one of the sessions entails completing 30 minutes of cognitive training session using the application. A ratio of completion will be calculated using the number of sessions completed over the total amount of sessions possible.

SECONDARY OUTCOMES:
Change in Corsi Task performance from baseline to 4 weeks | At baseline; Immediately after the 4-week study
  Visuospatial working memory will be measured with a modified Corsi Task, a collection of 4 types of tasks (i.e. classic - blocks, simple, complex, sequencing) that are customizable where an experimenter can select which task mode, stimulus type, and algorithm they want to use. In all versions of the task, the participant is shown instructions and then practices the task. Corsi Blocks Classic: The participant first completes Corsi Blocks Forward (tap in same order), followed by Corsi Blocks Reverse (tap in reverse order). The Corsi Blocks Forward task is split into two parts: the first is a method of limits to find the participants threshold, whereas the second provides additional trials around that threshold. Complex Corsi: Combines Simple Corsi with a secondary sorting task in between each trial. In the sorting task, the participant must drag a dog to a bone or a monkey to a banana. The location of the bone and banana are randomized to prevent mnemonic strategies like chunking.
Change in Letter-Number Task performance from baseline to 4 weeks | At baseline; Immediately after the 4-week study
  In the Letter-Number task, working memory will be assessed. Participants are presented with a mixed order of letters and numbers, which they must remember and sort them numerically and alphabetically. For example, the sequence 'H8T3K5' would be sorted into '358' and 'HKT'. The mixed orders of letter and numbers ranges from 2 to 15. After a short tutorial, the participant practices the task and must get three out of the five trials correct to proceed to the test. The Letter Number Task is split into two parts: The first is a method of limits to find the participants threshold, whereas the second provides additional trials around that threshold. Characters that could be confused with other letters or numbers are excluded (0, I, O, U, X). Moreover, a given sequence does not include any of the characters in the previous trial and it does not contain consecutive numbers and letters.
Change in N-Back Task performance from baseline to 4 weeks | At baseline; Immediately after the 4-week study
  In the N-Back task, working memory will be assessed. Participants are presented with a consecutive stream of pictures, and the objective is to tap on the pictures that match those presented N items earlier. Higher levels of N levels increase WM load and make the task more difficult. All participants complete 1-back (Figure 4), 2-back, and 3-back (in that order). Before each level starts, there is a practice session consisting of 10 trials during which performance feedback is provided. The test phase for each N-level consists of 30 trials with 9 targets. Progression to 4-back (and beyond) is allowed if the participant made no more than 2 errors on the previous level. Stimuli are presented for 2500 ms (participant can respond during this period) with an ISI of 500 ms.
Change in Cancellation Task performance from baseline to 4 weeks | At baseline; Immediately after the 4-week study
  The Cancellation Task is a timed, tablet-based test of selective attention and inhibitory control, akin to D2 (Brickenkamp & Zilmer, 1998). There are two versions that can be used interchangeably: Cancellation Letters and Cancellation Pictures. Cancellation - Letters resembles the D2 in that it consists of similar stimuli: characters "d" and "p" with one to four dashes, arranged either individually or in pairs above or below the letters. For Letters, the participant must scan the items from left to right and select all "d"s with two dashes (targets). In Cancellation - Pictures, letters are replaced with pictures of dogs and monkeys, some of which are rotated along the vertical axis or are presented upside down. For Pictures, the participant must select the upright dog (tail on the left) and the upside-down monkey (tail on right) separately in single blocks and together in a mixed block.
Change in Flanker Task performance from baseline to 4 weeks | At baseline; Immediately after the 4-week study
  The Flanker Task tests selective attention and inhibitory control. Participants are presented with a row of arrows and are asked whether the centrally presented arrow is pointing either to the left or to the right. In the congruent trials, the non-target arrows point in the same direction as the target arrow and in the incongruent trials they point in the opposite direction. The stimuli are presented in a pseudo-random order in which neither the trial type nor the trial direction can repeat more than three times in a row. Each condition is presented 12 times resulting in 48 total trials. The row of arrows is presented for 500ms with a 500ms break. The location of the row is randomly jittered so that it appears in one of 9 possible locations to prevent participants from fixating their gaze on the location of the central arrow. The user has 15 seconds to choose a response from the moment a trial is presented. Participants should respond as quickly and accurately as possible.
Change in Rule Switch Task performance from baseline to 4 weeks | At baseline; Immediately after the 4-week study
  The Rule Switch Task is a tablet-based measure of inhibitory control modeled after standard rule switching tasks such as the NIH Examiner (Kramer et al, 2014). In this task, participants must match the stimulus at the top of the screen (either a red or blue circle or square) by selecting one of the buttons (i.e., a red square or blue circle). Participants are instructed to classify the shape by one of two rules, either shape or color. There are 24 color trials and 24 shape trials, half of one shape and half of the other, for a total of 48 trials. There are three variables: shape, color and trial type. The three variables are pseudo-randomly intermixed so that any subset of 5 consecutive trials cannot have one of those traits in common across all 5 trials (no more than 4 trials in a row can share any of the three variable traits in common). There is also a switch rule in that there need to be a minimum of two trials of the same type before switching to a different trial type.
Experience with walking regimen and cognitive training | Immediately after the 4-week study
  Assessed by semi-structured interviews and will include: participants' satisfaction with the app and/or walking regime; perceived benefits of cognitive training and/or walking; and barriers to engaging with the app and/or walking regime.

OTHER OUTCOMES:
Executive functioning | At baseline; Immediately after the 4-week study
  Assessed using the Behavior Rating Inventory of Executive Function for Adults (BRIEF-A).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah J Salvy, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States